CLINICAL TRIAL: NCT04759157
Title: A Novel Couples- Based Sleep Health Intervention For Older Adults With Obstructive Sleep Apnea: Implications for Alzheimer's Disease Risk And Healthy Aging
Brief Title: We-PAP: A Couples-based Intervention for Sleep Apnea
Acronym: We-PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH); RAND (Other)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00135927; 1R21AG067183-01A1 (NIH)
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This is a dyadic study. Couples are randomly assigned as a dyad.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcomes assessors will not have knowledge of the randomization table. Participants will be reminded to not to tell the outcomes assessors their group. Only the statistician and interventionist will be aware of the group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Couples-based treatment- Patient (Experimental): Participants will attend 3, sessions (75, 50, 50 min) over video with a study therapist to discuss education about OSA and CPAP, strategies adjust to CPAP as a couple and techniques to improve sleep health.
  Interventions: Behavioral: Couples-based treatment
- Couples-based treatment- Partner (Experimental): Participants will attend 3, sessions (75, 50, 50 min) over video with a study therapist to discuss education about OSA and CPAP, strategies adjust to CPAP as a couple and techniques to improve sleep health.
  Interventions: Behavioral: Couples-based treatment
- Information Control- Patient (Active Comparator): Participants will receive treatment as usual and also standardized information about OSA and CPAP.
  Interventions: Other: Standardized education
- Information Control- Partner (Active Comparator): Participants will receive treatment as usual and also standardized information about OSA and CPAP.
  Interventions: Other: Standardized education

INTERVENTIONS:
Behavioral: Couples-based treatment — Couples will attend 3, video based sessions for couples-based treatment
  Arms: Couples-based treatment- Partner; Couples-based treatment- Patient
Other: Standardized education — Patients will receive standardized educational materials
  Arms: Information Control- Partner; Information Control- Patient

SUMMARY:
The purpose of this study is to develop, refine and evaluate the feasibility of a novel couples-based intervention to improve adherence for patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
This study will develop and test a novel couples-based intervention for the treatment of OSA and sleep health among older couples. The focus of this study is patient who are starting CPAP treatment and their partners. Couples will be randomized to a 3-session sleep health intervention delivered via telehealth or to standard educational support for CPAP. The intervention is based on a transdiagnostic model of sleep and circadian disorders (TransS-C) and rooted in the idea that older adults with OSA are often also having other sleep problems, and that OSA is best treated in the couples context.

ELIGIBILITY:
Inclusion Criteria:

Patient and partner inclusion criteria:

1. Age >=50
2. Access to cellular (active data plan) or Wi-Fi, in order to complete the telehealth intervention.

Patients inclusion criteria:

1. Diagnosed with OSA (AHI>10 or AHI>5 with impairment) and intend to start PAP treatment
2. PAP naïve or non-use of PAP for at least 3 years
3. Married or cohabiting with a romantic partner for >1 year
4. Able to read/write English.

Partner inclusion criteria:

1. Able to read/write English
2. PROMIS sleep disturbance score >55 in either patient or partner, or desire to improve sleep.

Exclusion Criteria:

Patient only exclusion criteria:

1. Concomitant OSA treatments (bariatric surgery planned in the next 3 months or bariatric surgery in the past year, ear nose and throat surgery for sleep apnea occurring in the 3 months before or planning for within the study period).

Exclusion criteria for both patient and partner include the following:

1. High risk or presence of moderate to severe comorbid sleep disorders (i.e., restless legs syndrome)
2. History of cognitive or neurological disorders (e.g., dementia, Parkinson's, Multiple Sclerosis)
3. Presence of major psychiatric disorders (e.g., schizophrenia, bipolar disorder), alcohol abuse reported on the Audit-C (score >4 for men, >3 for women), drug use (NIDA-Modified ASSIST score >3)
4. Unstable or serious medical illness that would interfere with participation (cancer, renal disease on dialysis, moderate to severe COPD)
5. Use of ASV, VPAP or supplemental oxygen
6. Overnight work > 1x per month
7. Pregnancy/ desire to become pregnant in the study period
8. Current participation in behavioral sleep treatment (e.g., CBT-I) or completion of CBT-I in the past 3 years
9. Concurrent participation in another clinical trial
10. Caregiving for an infant < 2 years old or adult who requires overnight assistance.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 1 year of completion of the study, will be available for 3 years.
Access Criteria: Written request to the PI

REFERENCES:
- [Derived] Baron KG, Gilles A, Sundar KM, Baucom BRW, Duff K, Troxel W. Rationale and study protocol for We-PAP: a randomized pilot/feasibility trial of a couples-based intervention to promote PAP adherence and sleep health compared to an educational control. Pilot Feasibility Stud. 2022 Aug 6;8(1):171. doi: 10.1186/s40814-022-01089-x. PMID 35933417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 2021 to October 2023 from the University of Utah Sleep Wake Center among patients who were undergoing sleep apnea testing (polysomnography and home sleep testing) for suspected sleep apnea.
  84 participants were consented and 74 continued to baseline assessment. A total of 10 individuals (5 couples) did not complete baseline for the following reason: 4 couples became ineligible (did not start PAP, started oxygen), 1 couple did not complete baseline.
Pre-assignment Details: Participants were recruited if they were planning to begin PAP treatment for obstructive sleep apnea.
Groups:
- Couples Based Treatment- Partner: Participants will attend 3, sessions (75, 50, 50 min) over video with a study therapist to discuss education about OSA and CPAP, strategies adjust to CPAP as a couple and techniques to improve sleep health.
  Couples-based treatment: Couples will attend 3, video based sessions for couples-based treatment
- Information Control- Patient; Information Control- Partner: Treatment as usual plus standardized educational materials
Period: Overall Study
Arm/Group | Couples-based Treatment- Patient | Couples Based Treatment- Partner | Information Control- Patient | Information Control- Partner
Started | 20 | 20 | 17 | 17
Completed | 20 | 20 | 17 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 84 individuals (42 couples) initially consented and 74 individuals (37) completed baseline assessments. A total of 10 participants (5 couples) were removed or declined to continue to baseline (4 couples became inelgibile and 1 declined)
Groups:
- Standard Information Control- Patient; Standard Information Control- Partner: Participants will receive treatment as usual and also standardized information about OSA and CPAP.
  Standardized education: Patients will receive standardized educational materials
- Total: Total of all reporting groups
Arm/Group | Couples-based Treatment- Patient | Couples-based Treatment- Partner | Standard Information Control- Patient | Standard Information Control- Partner | Total
Number analyzed (Participants) | 20 | 20 | 17 | 17 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 7 | 9 | 10 | 39
  >=65 years | 7 | 13 | 8 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data from 5 couples were removed from the analyses for the following reasons: Machine taken away before 3 months (n=2), random responding (n=1), cognitive impairment (n=1)
  years | 62.2 (7.4) | 59.9 (7.7) | 66.1 (8.8) | 64.3 (11.6) | 63.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data from 5 couples were removed from the analyses for the following reasons: Machine taken away before 3 months (n=2), random responding (n=1), cognitive impairment (n=1)
  Participants
    Female | 9 | 11 | 8 | 9 | 37
    Male | 11 | 9 | 9 | 8 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 18 | 16 | 16 | 15 | 65
  Unknown or Not Reported | 1 | 3 | 0 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 2 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 18 | 18 | 16 | 13 | 65
  More than one race | 2 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 17 | 17 | 74

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility
Description: Defined as the ability to achieve the recruitment goals of the study, to recruit approximately 3-4 couples per month over the study period (12 months)
Time Frame: study duration
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Patients recently diagnosed with obstructive sleep apnea (pre-randomization)
- Partners: Partners of patients recently diagnosed with obstructive sleep apnea (OSA), pre-randomization
Arm/Group | Patients | Partners
Number analyzed (Participants) | 42 | 42
Participants | 42 | 42

2. Secondary Outcome: Percentage of Days With PAP Use of 4 Hours or More
Description: The primary efficacy measure for this pilot trial was the percentage of days that patients used CPAP for 4 hours or more over the first 3 months. This 4 hour cutoff was selected becasue it is the minimum usage defined by Medicare and other insurance companies. We obtained patients' CPAP usage by downloading data from their machine using a remote dashboard. Data are only available for patients because partners were not using the treatment. This variable is defined as a proportion, calculated as the number of days with CPAP usage of 4 hours or more divided by the total number of days collected in the 3 month recording period. Scores can range from 0 (no days with use to 1, indicating all days with use of 4 hours or more).
Time Frame: 3 months
Population: Patients who had their PAP machine removed were given a zero at 3 months (n=2 patients)
Measure: Mean (Standard Deviation); unit: proportion of nights with CPAP >=4h
Arm/Group | Couples-based Treatment- Patient | Standard Information Control- Patient
Number analyzed (Participants) | 20 | 17
proportion of nights with CPAP >=4h | .73 (.08) | .72 (.07)
Statistical Analysis 1: Comparison: Couples-based Treatment- Patient vs Standard Information Control- Patient; Test type: Superiority; p = .30, mixed model

3. Secondary Outcome: Self-reported Sleep Disturbance
Description: Patient sleep quality on the Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance scale, 8 item, version 8b. Models evaluated change from baseline to 3 months. Raw are converted to t-scores, with a range of 28.9-76.5, a mean of 50 and a SD of 10. Higher scores indicate poorer sleep subjective quality.
Time Frame: 3 months
Population: Baseline PROMIS sleep quality data are missing for this variable for one couple in the intervention group and one couple in the control group
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Couples-based Treatment- Patient: Couples-based sleep health intervention
- Couples-based Treatment- Partner: Couples-based sleep-health intervention
- Standard Information Control- Patient; Standard Information Control- Partner: Information plus one follow-up phone call
Arm/Group | Couples-based Treatment- Patient | Couples-based Treatment- Partner | Standard Information Control- Patient | Standard Information Control- Partner
Number analyzed (Participants) | 20 | 20 | 17 | 17
t-score
  Baseline: number analyzed (Participants) | 19 | 19 | 16 | 16
  Baseline | 55.3 (6.8) | 50.6 (5.7) | 56.7 (7.8) | 48.6 (6.4)
  3 months | 49.6 (5.9) | 48.3 (6.3) | 51 (6.1) | 48.7 (6.9)
Statistical Analysis 1: Comparison: Couples-based Treatment- Patient vs Couples-based Treatment- Partner vs Standard Information Control- Patient vs Standard Information Control- Partner; We conducted multilevel models evaluating sleep disturbance score by assessment, group and patient versus partner status; Test type: Superiority; p = .206, Mixed Models Analysis; Mean Difference (Net) = -2.6, 95% CI 2-sided [-6.63 to 1.43], Standard Error of Mean 2.05 — This estimate is comparing intervention to control from baseline to 3 month for both patients and partners

4. Other Pre Specified Outcome: Intervention Completion
Description: Percentage of participants who completed the intervention sessions: 3 sessions for the couples-based treatment group and 1 handout and phone call for the information control group
Time Frame: intervention period, 1 month
Population: 100% of participants completed the planned intervention for their assigned group.
Measure: Count of Participants; unit: Participants
Arm/Group | Couples-based Treatment- Patient | Couples Based Treatment- Partner | Information Control- Patient | Information Control- Partner
Number analyzed (Participants) | 20 | 20 | 17 | 17
Participants | 20 | 20 | 17 | 17

5. Other Pre Specified Outcome: Retention
Description: We defined retention as the number of participants completing the 3 month follow-up. Our goal was to acheive at least 85% retention.
Time Frame: 3 months
Population: We acheived 100% retention, with all participants completing the 3 month follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Couples-based Treatment- Patient | Couples Based Treatment- Partner | Information Control- Patient | Information Control- Partner
Number analyzed (Participants) | 20 | 20 | 17 | 17
Participants | 20 | 20 | 17 | 17

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse reports were collected if reported by the participants in intervention sessions or assessment visits.
Groups:
- Standard Information Control- Patient; Standard Information Control- Partner: Standardized education: Patients will receive standardized educational materials plus one phone call
Arm/Group | Couples-based Treatment- Patient | Couples-based Treatment- Partner | Standard Information Control- Patient | Standard Information Control- Partner
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Limitations include: small sample size, enrollment at a single academic sleep center, primarily White sample with high educational attainment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT04759157/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04759157/SAP_001.pdf
  • Informed Consent Form (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT04759157/ICF_002.pdf